CLINICAL TRIAL: NCT04908280
Title: Exploratory Study of Ruxolitinib Cream for the Treatment of Discoid Lupus Erythematosus
Brief Title: Study of Ruxolitinib Cream for the Treatment of Discoid Lupus Erythematosus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Principal Investigator, Christopher T Richardson MD, PhD, Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00006186
Record Dates: First submitted 2021-05-26; First posted 2021-06-01 (Actual); Results first posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Discoid Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Discoid | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Discoid lupus erythematosus (Experimental): Patients with discoid lupus erythematosus will be given ruxolitinib cream to be used twice daily for 12 weeks.
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — 1.5% cream; Ruxolitinib cream will be applied topically twice daily to areas with active lesions.

SUMMARY:
The purpose of this study is to assess the potential efficacy of topical ruxolitinib for the treatment of discoid lupus erythematosus (DLE)

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and comply with the protocol and provide informed consent.
* Speaks English.
* Age ≥ 18 years.
* Clinical diagnosis of discoid lupus as assessed by the PI.
* At least one active (inflamed) discoid lesion with an IGA score of ≥ 3 and with a diameter ≥ 1cm at screening and baseline. Two lesions with equal scores will be necessary if consenting to pre-and post-treatment biopsies.
* Maximum body surface area of 20%.

Exclusion Criteria:

* Unwillingness or inability to complete informed consent process or comply with the study protocol.
* Pregnant or breast-feeding women, or women planning to become pregnant or breastfeed during the study.
* History of coagulopathy, pulmonary embolism or deep venous thrombosis.
* History of cutaneous squamous cell carcinoma localized to the treatment area.
* Serum creatinine > 1.5 mg/dL, or alanine aminotransferase or aspartate aminotransferase > 1.5 × upper limit of normal.
* Other dermatologic disease besides discoid lupus whose presence or treatments could complicate assessments.
* Other diseases besides dermatologic disorders whose treatment could complicate assessments. Subjects with systemic lupus erythematosus are permitted as long as they do not have unstable disease and meet all other criteria, including the exclusion criteria for systemic immunosuppressive or immunomodulating drugs (below).
* Topical treatments for discoid lupus within 2 weeks of Visit 2.
* Systemic immunosuppressive or immunomodulating drugs (e.g. oral or injectable corticosteroids, methotrexate, cyclosporine, mycophenolate mofetil, azathioprine) other than antimalarials (hydroxychloroquine, chloroquine, quinacrine) within 4 weeks or 5 half-lives of Visit 2 (whichever is longer).
* Potent systemic cytochrome P450 3A4 inhibitors or fluconazole within 2 weeks or 5 half-lives, whichever is longer, before Visit 2 (topical agents with limited systemic availability are permitted).
* Prior use of JAK inhibitors, systemic or topical, within the last 12 months.
* Ultraviolet (UV) therapy or tanning within 2 weeks prior to Visit 2 or during the duration of the treatment period.
* Any systemic or local infection that, in the opinion of the investigator, may compromise the safety of the subject or complicate assessments.
* Subjects allergic to lidocaine or with a history of keloids will not be allowed to provide an optional skin biopsy, but will be eligible for the remainder of the study.
* Electrocardiogram (ECG) changes on baseline screening consistent with high risk for a major adverse cardiovascular event (MACE).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-05-04 (Actual); Primary Completion 2024-03-04 (Actual); Study Completion 2024-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher T Richardson, MD, PhD, Principal Investigator — University of Rochester
Locations (1):
- UR Medicine Dermatology College Town, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Discoid Lupus Erythematosus
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Discoid Lupus Erythematosus
Number analyzed (Participants) | 10
Age, Continuous [Mean (Full Range); unit: years] | 49.9 [21 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10
Mean severity of disease as measured by the Investigator's Global Assessment [Mean (Standard Deviation); unit: score on a scale] — The Investigator's Global Assessment will be performed at study visits 2-6. The IGA is an instrument to rate the severity of the subject's global disease. This IGA is comprised of a 5-point scale of disease activity ranging from 0 to 4 as follows: 0: "clear," no erythema or scale
  1. "almost clear," pink erythema without scale
  2. "mild," pink erythema with scale
  3. "moderate," red erythema with scale
  4. "severe," purple/violaceous or hemorrhagic/crusted erythema OR hypertrophic/ verrucous scale
  Range of scores are 0-4 with higher scores indicating worse outcome.
  score on a scale | 3.0 (0)
Mean itch symptoms [Mean (Standard Deviation); unit: score on a scale] — Subjects will maintain a symptom diary every day for 12 weeks. Specifically, subjects will rate pain and itch separately using a numeric rating scale (NRS) and the questions below. Symptom diaries will be reviewed at study visits 2-6. "On a scale of "no itch" (0) to "worst imaginable itch" (10), how was your worst itch in the 24 hours?"
  Scores will range from 0-10 with higher scores indicating worse outcome.
  score on a scale | 2.8 (4.12)
Mean pain symptoms [Mean (Standard Deviation); unit: score on a scale] — Subjects will maintain a symptom diary every day for 12 weeks. Specifically, subjects will rate pain and itch separately using a numeric rating scale (NRS) and the questions below. Symptom diaries will be reviewed at study visits 2-6.
  "On a scale of "no skin pain" (0) to "worst imaginable skin pain" (10), how was your worst skin pain in the 24 hours?"
  Scores will range from 0-10 with higher scores indicating worse outcome.
  score on a scale | 1.2 (3.16)

OUTCOME MEASURES:

1. Primary Outcome: Mean Severity of Disease as Measured by the Investigator's Global Assessment
Description: The Investigator's Global Assessment will be performed at study visits 2-6. The IGA is an instrument to rate the severity of the subject's global disease. This IGA is comprised of a 5-point scale of disease activity ranging from 0 to 4 as follows: 0: "clear," no erythema or scale
  1. "almost clear," pink erythema without scale
  2. "mild," pink erythema with scale
  3. "moderate," red erythema with scale
  4. "severe," purple/violaceous or hemorrhagic/crusted erythema OR hypertrophic/ verrucous scale
  Range of scores are 0-4 with higher scores indicating worse outcome.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Discoid Lupus Erythematosus
Number analyzed (Participants) | 10
score on a scale | 1.4 (0.84)

2. Secondary Outcome: Mean Percentage Change in Disease Activity as Measured by the Cutaneous Lupus Area and Severity Index-A (CLASI)
Description: The Cutaneous Lupus Area and Severity Index (CLASI) will be performed at study visits 2-6. This is a validated measurement instrument designed for use in clinical trials to assess disease activity and damage in subjects with cutaneous lupus. The CLASI is comprised of two parts, CLASI-A that measures disease activity (erythema and scale), and CLASI-D that measures disease damage (pigmentation and scarring).
  CLASI-A scores range from 0 to 70 with higher scores indicating worse outcomes.
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: percentage of change in disease activity
Arm/Group | Discoid Lupus Erythematosus
Number analyzed (Participants) | 10
percentage of change in disease activity | -30.2 (25.8)
Statistical Analysis 1: Comparison: Discoid Lupus Erythematosus; Test type: Superiority; p = 0.0308, ANOVA

3. Secondary Outcome: Mean Change in Itch Symptoms
Description: Subjects will maintain a symptom diary every day for 12 weeks. Specifically, subjects will rate pain and itch separately using a numeric rating scale (NRS) and the questions below. Symptom diaries will be reviewed at study visits 2-6. "On a scale of "no itch" (0) to "worst imaginable itch" (10), how was your worst itch in the 24 hours?"
  Scores will range from 0-10 with higher scores indicating worse outcome.
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Discoid Lupus Erythematosus
Number analyzed (Participants) | 10
score on a scale | 0.67 (2.00)

4. Secondary Outcome: Mean Change in Pain Symptoms
Description: Subjects will maintain a symptom diary every day for 12 weeks. Specifically, subjects will rate pain and itch separately using a numeric rating scale (NRS) and the questions below. Symptom diaries will be reviewed at study visits 2-6.
  "On a scale of "no skin pain" (0) to "worst imaginable skin pain" (10), how was your worst skin pain in the 24 hours?"
  Scores will range from 0-10 with higher scores indicating worse outcome.
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Discoid Lupus Erythematosus
Number analyzed (Participants) | 10
score on a scale | 0.67 (2.00)

5. Secondary Outcome: Mean Change in Melanin Index Score
Description: Photographs of all discoid lesions will be taken at baseline and week 12. The Haiku app will be used to directly load photos into the secure Epic medical record system. Images will be extracted from Epic, and analyzed. In brief, a melanin index (MI) will be generated for each lesion using Image J software analysis. The measurement will be a ratio comparing the pigmentation of the lesion to non-lesion skin. The analysis uses perilesional skin to normalize the photograph.
  Measurements will range from 0 to 10. Scores further from a score of 1 will indicate more severe outcomes.
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: photographs
Arm/Group | Discoid Lupus Erythematosus
Number analyzed (Participants) | 10
Number analyzed (photographs) | 60
score on a scale
  baseline | 2.28 (1.18)
  12 weeks | 2.73 (2.36)

6. Secondary Outcome: Mean Change in Erythema Index Score
Description: Photographs of all discoid lesions will be taken at baseline and week 12. The Haiku app will be used to directly load photos into the secure Epic medical record system. Images will be extracted from Epic, and analyzed. In brief, an erythema index (EI) will be generated for each lesion using Image J software analysis. The measurement will be a ratio comparing the erythema of the lesion to non-lesion skin. The analysis uses perilesional skin to normalize the photograph.
  Measurements will range from 0 to 10. Scores further from a score of 1 will indicate more severe outcomes.
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: photographs
Arm/Group | Discoid Lupus Erythematosus
Number analyzed (Participants) | 10
Number analyzed (photographs) | 60
score on a scale
  baseline | 1.87 (0.74)
  12 weeks | 1.18 (0.18)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Discoid Lupus Erythematosus
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-06): https://cdn.clinicaltrials.gov/large-docs/80/NCT04908280/Prot_SAP_000.pdf
  • Informed Consent Form (2023-10-03): https://cdn.clinicaltrials.gov/large-docs/80/NCT04908280/ICF_001.pdf